CLINICAL TRIAL: NCT01359111
Title: Phase I Performance and Safety Evaluation of an Intradermal Delivery Device
Brief Title: Performance and Safety Evaluation of an Intradermal Delivery Device
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PATH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HS 563
Record Dates: First submitted 2011-05-02; First posted 2011-05-24 (Estimated); Results first posted 2012-05-11 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Injections, Intradermal
Keywords: Intradermal injections; Vaccination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: PATH ID Adapter — Intradermal delivery device which fits on the end of a syringe to limit the depth and angle of needle penetration into the skin.

SUMMARY:
The purpose of this study is to evaluate whether an investigational vaccine delivery device (the ID adapter) can safely and precisely inject liquid into the intradermal layer of the skin.

ELIGIBILITY:
Inclusion Criteria:

* Female and male participants ages 18 to 55 years.
* Healthy enough to participate in the clinical trial per site investigator assessment.
* Healthy skin on the upper deltoid region of both arms.
* Able to provide signed informed consent and understand study procedures per ICH/GCP guidelines.
* Literate in English.
* Available by telephone 48 hours after the study visit.

Exclusion Criteria:

* Skin abnormalities on upper deltoid region of either arm (scars, rash, infection) or other skin conditions that would interfere with the ability to visualize an intradermal injection in the opinion of the investigator.
* Unable to understand the study purpose or procedures.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Klaff, MD, PhD, Principal Investigator — Rainier Clinical Research Center
Locations (1):
- Rainier Clinical Research Center, Renton, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intradermal Adapter: Saline injection with intradermal adapter
Period: Overall Study
Arm/Group | Intradermal Adapter
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intradermal Adapter
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 35.4 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Injections Delivered to the Intradermal Layer of the Skin
Description: The proportion of saline injections via the ID Adapter resulting in delivery to the intradermal layer of the skin will be assessed by visualization of intradermal wheals with diameters ≥ 5mm, the volume of liquid injected, and confirmation of delivery to the intradermal layer by ultrasound.
Time Frame: 1 day
Measure: Number; unit: percentage of injections
Units Other Than Participants: injections
Arm/Group | Intradermal Adapter
Number analyzed (Participants) | 20
Number analyzed (injections) | 40
percentage of injections | 1

2. Secondary Outcome: Proportion of Participants With Safety Events
Description: The proportion of participants with safety events will be calculated for events occurring within 30 minutes and within 48 hours of injection.
Time Frame: 2 days
Measure: Number; unit: percentage of participants
Arm/Group | Intradermal Adapter
Number analyzed (Participants) | 20
percentage of participants | 0.25

3. Secondary Outcome: Proportion of Injections Administered With Needle Bevel up and Needle Bevel Down Delivered to the Intradermal Layer of the Skin.
Description: The proportion of saline injections administered with the ID Adapter with needle bevel oriented up and needle bevel oriented down resulting in delivery to the intradermal layer of the skin. This will be assessed by visualization of intradermal wheals with diameters ≥ 5mm, the volume of liquid injected, and confirmation of delivery to the intradermal layer by ultrasound.
Time Frame: 1 day
Measure: Number; unit: percentage of injections
Units Other Than Participants: injections
Groups:
- Bevel Up: Saline injection with intradermal adapter used with needle bevel oriented up relative to the surface of the skin
- Bevel Down: Saline injection with intradermal adapter used with needle bevel oriented down relative to the surface of the skin
Arm/Group | Bevel Up | Bevel Down
Number analyzed (Participants) | 20 | 20
Number analyzed (injections) | 20 | 20
percentage of injections | 1 | 1

ADVERSE EVENTS:
Time Frame: 2 days
Arm/Group | Intradermal Adapter
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 5/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intradermal Adapter (N=20)
Abrasion (Skin and subcutaneous tissue disorders) | 5 (5) — Superficial abrasion of skin caused by the needle scratching the skin as the intradermal adapter and syringe moved horizontally along the surface of the skin prior to initial skin penetration

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No